CLINICAL TRIAL: NCT02960802
Title: Kidney Transplantation and Renal and Myocardial Perfusion
Acronym: Transkidney
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Johanna Paivarinta, MD, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T257/2016
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Kidney Transplant Failure
Keywords: kidney transplant; renal blood flow
MeSH Terms: interventions — Kidney Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- kidney transplant patient (Active Comparator): kidney transplantation is intervention
  Interventions: Procedure: kidney transplantation
- healthy control (No Intervention): no intervention

INTERVENTIONS:
Procedure: kidney transplantation
  Other Names: transplant
  Arms: kidney transplant patient

SUMMARY:
The cardiovascular morbidity and mortality is significantly higher in chronic kidney disease (CKD) patients, especially in dialysis patients, than in normal population. The increased risk of cardiovascular diseases is multifactorial.Endothelial dysfunction is one of the explanations for the poor outcome of kidney patients. The kidney transplantation seems to halt the progression of the cardiovascular morbidity.

Coronary flow reserve (CFR), the capacity of coronary vessels to dilate in response to vasoactive agent, is a marker of the endothelial dysfunction. It is reduced in renal impairment as well as in many preatherosclerotic states and coronary heart disease. The method of choice to evaluate CRF is positron emission tomography (PET). In kidney transplant patients CFR seems to be worse than in healthy controls but better than in dialysis patients. However, the evidence is scarce.

Renal flow reserve (RFR) is smaller than that of heart. RFR probably reflects endothelial function in the same way as CFR does. Declining RFR could perhaps be used to anticipate worsening kidney function especially in kidney transplant patients and be in favour for transplant biopsy.There are no studies of RFR in renal allograft patients.

The objectives of this study are to examine the effect of kidney transplantation on coronary flow reserve (CFR), the change of renal flow reserve (RFR) in kidney transplant patients during the first year after transplantation and assess the correlation between the change of renal blood flow / RFR and kidney biopsy findings in kidney transplant patients.

The first hypothesis of this study is that coronary flow reserve of transplant patients is better than that of dialysis patients but worse than that of healthy controls. The second hypothesis is that renal transplant perfusion reserve is better at one year than at three months after transplantation. The third hypothesis is that pathologic kidney biopsy findings correlate negatively with renal perfusion reserve.

DETAILED DESCRIPTION:
INTRODUCTION Cardiovascular morbidity and kidney impairment Patients with chronic kidney disease (CKD) have a high risk of cardiovascular events and that is already substantial in early stages of CKD. The pathophysiology of cardiovascular disease in CKD patients is poorly understood. In end stage renal disease sudden arrhythmic cardiac death rather than myocardial infarction due to atherosclerosis is the predominant cause of cardiovascular mortality. In uremia endothelial vasodilation is impaired. This may be one explanation for the high prevalence of cardiovascular disease in CKD.The renal transplantation reduces cardiovascular risk and improves the patient survival.

The traditional approaches for cardiac risk assessment like SPECT-MPI (single photon emission computed tomography-myocardial perfusion imaging) are perhaps not as liable in chronic kidney disease patients than in healthy population. Coronary angiography is invasive and may induce contrast nephropathy and deteriorating kidney function.

The coronary flow reserve (CFR) or myocardial flow reserve (MFR) is the magnitude of increase in coronary flow which is calculated assessing myocardial blood flow at rest (basal flow) and during pharmacological vasodilation and hyperemia.Myocardial blood flow (MBF) needs to dynamically adapt to the metabolic demand of the myocardium and it is controlled by coronary microvascular resistance. Microvascular dysfunction may be caused by different mechanisms, one of them is microvascular dysfunction.

CFR has been measured by transthoracic echocardiography(TTEC) as well as intracoronary Doppler echocardiography has been used to estimate CFR. However, blood velocity measurement in one coronary artery is not the same as quantification of myocardial blood flow.Magnetic resonance imaging (MRI) can be used to quantify myocardial blood flow as well but it is not safe in renal impairment because of the contrast agent gadolinium. In recent years PET has shown to be the modality of choice to measure myocardial blood flow (MBF). It is noninvasive and it is safe in renal impairment.

High prevalence of cardiovascular morbidity in CKD-patients is not only explained by large vessel atherosclerosis. It has been shown poor cardiac outcome in CKD-patients without obstructive coronary artery disease. The dysfunction of microvasculature may be one explanation in such circumstances.

Despite the evidence of the increased prevalence of coronary artery disease in CKD patients there are only a quite few studies of coronary flow reserve in this subgroup of patients, especially positron emission tomography (PET) studies.The results of these studies are controversial.

As kidney transplantation decreases the uremic effect on cardiovascular system it is likely that it has also an impact on CFR. Endothelial function seems to improve after renal transplantation.There are only four studies of kidney transplant patients and their coronary flow reserve. None of them is done with PET which is the modality of choice estimating myocardial blood flow. The total number of patients in all these studies is 107.

In all of the studies CFR is reduced in renal transplant patients compared to normal but not as much as in ESRD patients in dialysis.

Renal blood flow Renal blood flow (RBF) RBF is a combination of blood flow in renal arteries and small vessels in the same way as coronary blood flow is a combination of blood flow in coronary arteries and microvasculature in the myocardium. It is probable that renal perfusion and flow reserve are dependent on endothelial function in the same way as myocardial perfusion is. Clinical disorders, such as renovascular hypertension or kidney impairment , are shown to reduce RBF. The ability to measure accurately the renal blood flow may help us to understand renal disease mechanisms and possibly even focus the right therapy at the right time.

In clinical practice, RBF can be measured indirectly by para-aminohippuric acid (PAH) clearance. It can not be used in renal impairment because of the decreased tubular excretion. Furthermore, it gives only two-kidney value. Renograms give no quantitative measurement either and are not interpretable in chronic kidney disease. Computed tomography can not be used in renal impairment because of nephrotoxicity of contrast agents.

Magnetic resonance imaging (MRI) MRI with gadolinium based contrast agents is contraindicated especially in CKD patients with GFR<30 ml/min because the risk of nephrogenic systemic fibrosis (NSF). However, new functional MRI methods without the need for contrast agent have been introduced during the past decades. None of them show real kidney perfusion.

Positron emission tomography (PET) PET provides a method to estimate quantitative regional renal cortical blood flow noninvasively. Nitzsche et al. were the first to develop and report the quantitative estimation of RBF using dynamic PET with H(2)(15)O. Kudomi et al. have demonstrated the feasibility of measurement of RBF using PET with H(2)(15)O in humans (63).H(2)(15)O is convenient because of its short half-life (2 minutes).It allows repeated measures with short intervals of 15 minutes. Furthermore, H(2)(15)O is fully diffusible tracer without dependency on tubular function and it´s not nephrotoxic. Irradiation to patient is low.

Only two studies of renal perfusion with PET was found in literature. Koivuviita et al. studied the effect of revascularisation on renal artery stenosis on renal perfusion in patients with atherosclerotic renovascular disease (ARVD) using PET. The cortical renal perfusion was correlated with the degree of stenosis in the renal artery, but it did not increase after revascularization. The mean cortical renal perfusion value in healthy controls was significantly higher than in CKD-patients. Moreover, the RBF was lower in diabetic than non-diabetic ARVD patients.In a study of Alpert et al. there were 5 subjects with normal renal function and 10 with moderate to severe renal disease. In CKD group there were also 4 renal transplant patients. The RBF was significantly higher in healthy controls than in CKD group.

There is no renal perfusion study done by PET in kidney transplant patients. Renal flow reserve Renal flow reserve (RFR) is the capacity of the renal circulation to augment renal bloodflow. It is possible that endothelial dysfunction in renal microvasculature decreases RFR. Furthermore, the decreased RFR could be a sign of pathologic process in kidney parenchyma.

Beregi et al. has shown with combination of angiography and intravascular Doppler in pigs that RFR is less marked than CFR . Hollenberg et al studied renal vasomotion with scintigraphic xenon-technique. The increase of renal blood flow was 20-35% in normotensive patients. Phentolamine, acetylcholine and diltiazem were dosed in renal artery, teprotide intravenously and captopril orally at the dose of 10-25 mg.Manoharan et al.used intrarenal Doppler and angiography to estimate the vasodilatory capacity of renal microvasculature in normotensive and normoglycemic adults with normal kidney function. The normal renal flow reserve averaged 2. PAH clearance was used as method in a IgA nephropathy study of Coppo et al.. The influence of oral captopril 50 mg on PAH clearance and effective renal bloodflow (ERBF) in CKD patients with moderate renal impairment and in healthy controls was evaluated. The ERBF was increased significantly in both groups after captopril. The tendency of lower basal flow values in CKD group was seen compared to controls.

There are some studies done with PET to evaluate changes in renal blood flow. Juillard et al. demonstrated in a pig study that angiotensin II reduces RBF and dopamine increases it. They also estimated RBF with means of PET using H(2)(15)O before and after quinaprilat injection (10 mg) in eight men with hypertension and moderate CRF. Baseline ERPF were decreased significantly. PET-RBF increased significantly after quinaprilat injection. No RFR-studies are done in kidney transplant patients.

Renal flow reserve and kidney transplantation The slowly deteriorating renal transplant is still a major concern of nephrologists. Sequential biopsies may help to predict the subsequent developing allograft nephropathy but the procedure is highly invasive. Renal blood flow and renal flow reserve may be informative in predicting renal transplant function.However, there is neither study of renal blood flow reserve nor renal blood flow done with PET based methodology in kidney recipients.

STUDY DESIGN One part of this study is a prospective longitudinal follow-up study and the other part is a retrospective cohort study. The centres involved in this study are Turku University Hospital Nephrology department and Turku PET centre.

1. .CFR is measured with PET in kidney transplant patients with diabetes and without diabetes whose GFR is more than 30 - 45 ml/min. The kidney transplant age should be 3+/- 1 years (retrospective).
2. .CFR of the dialysis patients on the kidney waiting list is measured by PET during dialysis time and at one year after kidney transplantation(prospective). Half of the patients are peritoneal dialysis patients and half of them hemodialysis patients.
3. .RFR/RBF of the kidney transplant recipients is measured with PET during the third month after kidney transplantation and at one year after transplantation (prospective).
4. .RBF/RFR of kidney transplant patients with GRF more than 30-45 ml/min is measured with PET. The kidney transplant age should be 3+/-1 years (retrospective).
5. .Coronary flow reserve with PET and RFR/RBF of healthy controls are measured.

Description of the measurement of coronary flow reserve (CFR) The PET imaging will be performed after a 10-h overnight fast. Alcohol, smoking and caffeine are prohibited 3 days before assessment. Antihypertensive medication should be interrupted 3 days before examinations.

The subjects are positioned supine in the PET tomograph. A venous catheter is inserted in an antecubital vein for injection of oxygen-15-labeled water ([15O]H2O). Myocardial perfusion is measured both at rest and two minutes after the end of adenosine infusion. All PET data are corrected for dead time, decay and measured photon attenuation. Images are processed with the standard reconstruction algorithm.Regions of interest (ROIs) are drawn on the left ventricle (LV) myocardium on an average of four midventricular transaxial planes covering the septum, anterior wall, lateral wall and the whole LV myocardium. The left ventricular cavity ROI is drawn and used as the input function for determination of the LV time-activity curve. Regional myocardial perfusion (ml/g tissue per min) is calculated with a single compartment model.

Description of the measurement of renal blood flow (RBF)/renal flow reserve (RFR) The instructions and limitations for the subjects before the procedure are the same as above. A venous catheter is inserted in an antecubital vein for injection of oxygen-15-labeled water ([15O]H2O). Renal perfusion data is corrected for dead time, decay and measured photon attenuation. Images are processed with the standard reconstruction algorithm. Regions of interest (ROI) for the whole cortical region of the kidneys are drawn on a summed reconstructed image on an average of six coronal planes. For the calculation of renal perfusion from the PET study, the input function is is estimated using an average time activity curve (TAC) from descending aorta cavity ROIs drawn on average three planes. Renal perfusion images are generated from the reconstructed dynamic image and the obtained input function by a basis function method assuming a single-tissue compartment model. Enalapril will be used at the dose of 0,5 mg-1 mg intravenously. Dose of radiation is reported separately.

5.2 Number of subjects

1. New kidney transplant patients without diabetes N=10-20
2. New kidney transplant patients with diabetes I or II N=10-20
3. "Old" kidney transplant patients with type I diabetes N=15-30
4. "Old" kidney transplant patients without diabetes N=15-30
5. Healthy controls N = 10

For patient registries:

1. Quality assurance and data validation is done by Turku Finland PET center. Registry procedures concerning patient data are handled by Southwestern hospital district of Finland.
2. Patients are recruited from the area of Turku university hospital during standard policlinic visits and in dialysis. Data is collected via imaging as previously described and data is managed and analysed in PET center. PET center reports for adverse events as well.
3. Efficacy calculations can´t be done because of the small number of patients. There is about 10 kidney transplantations / year in the hospital area.
4. If data is missing, it is reported.
5. The statistical methods include correlation analyses and tests are chosen depending of the distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* dialysis patients who are on the kidney waiting list

Exclusion Criteria:

* diabetes, hypertension, coronary artery disease, cerebrovascular disease, universal atherosclerosis

In the retrospective part of the study, inclusion criteria:

* kidney transplant is 3+/-1years old
* GFR >30 ml/min Exclusion criteria
* manifest coronary artery disease, cerebrovascular disease, universal atherosclerosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
renal flow reserve of kidney transplant patients | one year
  renal flow reserve of kidney transplant patients is measured by PET-camera at 3 months and at one year after transplantation, unit is ml/ml (blood/renal tissue)
cardiac flow reserve of kidney transplant patients | supposed to be 1-3 years depending how quickly patient gets the transplant
  cardiac flow reserve is measured by PET-camera during dialysis time and at one year after transplantation, unit is ml/g

SECONDARY OUTCOMES:
the difference of cardiac flow reserve of kidney transplant patients who have been previously peritoneal dialysis or hemodialysis patients | supposed to be 1-3 years depending how quickly patient gets the transplant
  the cardiac flow reserve is measured by PET during dialysis and at one year after kidney transplantation, unit is ml/g

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Päivärinta, MD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No
Data is obtained via imaging (PET). The data includes perfusion values of kidneys and heart. The data will be available in the end of study period, 12/2022.

REFERENCES:
- [Result] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Result] Culleton BF, Larson MG, Wilson PW, Evans JC, Parfrey PS, Levy D. Cardiovascular disease and mortality in a community-based cohort with mild renal insufficiency. Kidney Int. 1999 Dec;56(6):2214-9. doi: 10.1046/j.1523-1755.1999.00773.x. PMID 10594797
- [Result] Morris ST, McMurray JJ, Rodger RS, Jardine AG. Impaired endothelium-dependent vasodilatation in uraemia. Nephrol Dial Transplant. 2000 Aug;15(8):1194-200. doi: 10.1093/ndt/15.8.1194. PMID 10910444
- [Result] Al-Mallah MH, Hachamovitch R, Dorbala S, Di Carli MF. Incremental prognostic value of myocardial perfusion imaging in patients referred to stress single-photon emission computed tomography with renal dysfunction. Circ Cardiovasc Imaging. 2009 Nov;2(6):429-36. doi: 10.1161/CIRCIMAGING.108.831164. Epub 2009 Sep 8. PMID 19920040
- [Result] Jerosch-Herold M, Wilke N, Stillman AE. Magnetic resonance quantification of the myocardial perfusion reserve with a Fermi function model for constrained deconvolution. Med Phys. 1998 Jan;25(1):73-84. doi: 10.1118/1.598163. PMID 9472829
- [Result] Dries DL, Exner DV, Domanski MJ, Greenberg B, Stevenson LW. The prognostic implications of renal insufficiency in asymptomatic and symptomatic patients with left ventricular systolic dysfunction. J Am Coll Cardiol. 2000 Mar 1;35(3):681-9. doi: 10.1016/s0735-1097(99)00608-7. PMID 10716471
- [Result] Palmer RM, Ferrige AG, Moncada S. Nitric oxide release accounts for the biological activity of endothelium-derived relaxing factor. Nature. 1987 Jun 11-17;327(6122):524-6. doi: 10.1038/327524a0. PMID 3495737
- [Result] Green MA, Hutchins GD. Positron emission tomography (PET) assessment of renal perfusion. Semin Nephrol. 2011 May;31(3):291-9. doi: 10.1016/j.semnephrol.2011.05.008. PMID 21784278
- [Result] Koivuviita N, Liukko K, Kudomi N, Oikonen V, Tertti R, Manner I, Vahlberg T, Nuutila P, Metsarinne K. The effect of revascularization of renal artery stenosis on renal perfusion in patients with atherosclerotic renovascular disease. Nephrol Dial Transplant. 2012 Oct;27(10):3843-8. doi: 10.1093/ndt/gfs301. Epub 2012 Jul 10. PMID 22785108
- [Result] Alpert NM, Rabito CA, Correia DJ, Babich JW, Littman BH, Tompkins RG, Rubin NT, Rubin RH, Fischman AJ. Mapping of local renal blood flow with PET and H(2)(15)O. J Nucl Med. 2002 Apr;43(4):470-5. PMID 11937589
- [Result] Beregi JP, Lahoche A, Willoteaux S, McFadden E, Bordet R, Gautier C, Etchrivi T. Renal artery vasomotion: in vivo assessment in the pig with intravascular Doppler. Fundam Clin Pharmacol. 1998;12(6):613-8. doi: 10.1111/j.1472-8206.1998.tb00994.x. PMID 9818293
- [Result] Hollenberg NK, Sandor T. Vasomotion of renal blood flow in essential hypertension. Oscillations in xenon transit. Hypertension. 1984 Jul-Aug;6(4):579-85. doi: 10.1161/01.hyp.6.4.579. PMID 6746087
- [Result] Manoharan G, Pijls NH, Lameire N, Verhamme K, Heyndrickx GR, Barbato E, Wijns W, Madaric J, Tielbeele X, Bartunek J, De Bruyne B. Assessment of renal flow and flow reserve in humans. J Am Coll Cardiol. 2006 Feb 7;47(3):620-5. doi: 10.1016/j.jacc.2005.08.071. Epub 2006 Jan 18. PMID 16458147
- [Result] Juillard L, Janier MF, Fouque D, Cinotti L, Maakel N, Le Bars D, Barthez PY, Pozet N, Laville M. Dynamic renal blood flow measurement by positron emission tomography in patients with CRF. Am J Kidney Dis. 2002 Nov;40(5):947-54. doi: 10.1053/ajkd.2002.36325. PMID 12407639
- [Result] Bosmans JL, Ysebaert DK, Verpooten GA. Chronic allograft nephropathy: what have we learned from protocol biopsies? Transplantation. 2008 Apr 15;85(7 Suppl):S38-41. doi: 10.1097/TP.0b013e318169c5d0. PMID 18401262
- See also: N Engl J Med. 2004 Sep 23;351(13):1296-305 — https://www.ncbi.nlm.nih.gov/pubmed/15385656
- See also: Kidney Int. 1999 Dec;56(6):2214-9. — https://www.ncbi.nlm.nih.gov/pubmed/10594797
- See also: Nephrol Dial Transplant. 2000 Aug;15(8):1194-200. — https://www.ncbi.nlm.nih.gov/pubmed/10910444
- See also: Circ Cardiovasc Imaging. 2009 Nov;2(6):429-36 — https://www.ncbi.nlm.nih.gov/pubmed/19920040
- See also: Med Phys. 1998 Jan;25(1):73-84 — https://www.ncbi.nlm.nih.gov/pubmed/9472829
- See also: J Am Coll Cardiol. 2000 Mar 1;35(3):681-9 — https://www.ncbi.nlm.nih.gov/pubmed/?term=dries+prognostic+implications+of+renal
- See also: Nature. 1987 Jun 11-17;327(6122):524-6. — https://www.ncbi.nlm.nih.gov/pubmed/3495737
- See also: Semin Nephrol. 2011 May;31(3):291-9 — https://www.ncbi.nlm.nih.gov/pubmed/21784278
- See also: Nephrol Dial Transplant. 2012 Oct;27(10):3843-8 — https://www.ncbi.nlm.nih.gov/pubmed/?term=koivuviita+liukko+the+effect+of+revascularisation
- See also: J Nucl Med. 2002 Apr;43(4):470-5. — https://www.ncbi.nlm.nih.gov/pubmed/?term=alpert+mapping+of+local+renal+blood+flow+with+pet
- See also: Fundam Clin Pharmacol. 1998;12(6):613-8. — https://www.ncbi.nlm.nih.gov/pubmed/?term=beregi+renal+artery+vasomotion+doppler
- See also: Hypertension. 1984 Jul-Aug;6(4):579-85 — https://www.ncbi.nlm.nih.gov/pubmed/6746087
- See also: J Am Coll Cardiol. 2006 Feb 7;47(3):620-5. — https://www.ncbi.nlm.nih.gov/pubmed/16458147
- See also: Am J Kidney Dis. 2002 Nov;40(5):947-54. — https://www.ncbi.nlm.nih.gov/pubmed/?term=juillard+dynamic+renal+blood+flow+amj+kidney+dis
- See also: Transplantation. 2008 Apr 15;85(7 Suppl):S38-41 — https://www.ncbi.nlm.nih.gov/pubmed/18401262